CLINICAL TRIAL: NCT02913170
Title: Nattokinase Supplementation and Hemostatic Factors
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Jong Ho Lee, Professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: NP_intervention
Record Dates: First submitted 2016-09-20; First posted 2016-09-23 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — nattokinase

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nattokinase group (Experimental): A nattokinase group composed of 50 individuals who consumed a 300mg nattokinase capsule (100mg of nattokinase and 200mg of maltodextrin) daily after meal.
  Interventions: Dietary Supplement: Nattokinase
- Placebo group (Placebo Comparator): A placebo group composed of 50 individuals who consumed a 300mg placebo capsule (300mg of maltodextrin) daily after meal.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nattokinase
  Arms: Nattokinase group
Dietary Supplement: Placebo
  Arms: Placebo group

SUMMARY:
The aim of this study is to examine the effects of nattokinase supplementation on hemostatic factors in nondiabetic and hypercholesterolemic subjects. Collagen-epinephrine closure time, prothrombin time, activated partial thromboplastin time, fibrinogen levels, and lipid profiles were measured at baseline and at 8-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 69 years
* Hypercholesterolemia (200mg/dL ≤ serum cholesterol ≤ 280mg/dL)
* Nondiabetic (fasting blood glucose < 126mg/dL and 2-hour blood glucose < 200mg/dL)

Exclusion Criteria:

* Use of any medication or supplements
* Diagnosis of dyslipidemia, diabetes mellitus, hypertension, liver disease, renal disease, cardiovascular disease, pancreatitis, cancer, or any life-threatening illness that required regular medical treatment
* Women who were pregnant, breastfeeding or intending to become pregnant during the study period
* Drug or alcohol abuse

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Collagen-epinephrine closure time at baseline | baseline
Collagen-epinephrine closure time at 8-week follow-up | 8-week follow-up

SECONDARY OUTCOMES:
Prothrombin time at baseline | baseline
Prothrombin time at 8-week follow-up | 8-week follow-up
  second
Activated partial thromboplastin time at baseline | baseline
Activated partial thromboplastin time at 8-week follow-up | 8-week follow-up
Fibrinogen concentration at baseline | baseline
  mg/dL
Fibrinogen concentration at 8-week follow-up | 8-week follow-up
  mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Jong Ho Lee, Ph.D., Principal Investigator — Yonsei University
Locations (1):
- Laboratory of Clinical Nutrigenetics/Nutrigenomics, Yonsei University., Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No